CLINICAL TRIAL: NCT03654781
Title: Periodontal Tedavinin Helikobakter Pilori Eradikasyon ve Rekürrensine Katkısının İncelenmesi
Brief Title: Impact of Periodontal Treatment on Gastric Helicobacter Pylori Eradication
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ayla Öztürk, Associate Professor, Ondokuz Mayıs University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OndokusMU1; OMUetik 2009/95 (Other: Ondokuz Mayıs University)
Record Dates: First submitted 2018-06-10; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: periodontal treatment; Initial periodontal therapy; H. pylori

STUDY DESIGN:
Intervention Model Description: Participants with positive for both for H. pylori in gastric biopsy specimens and dental plaque samples by histologic examination with immunostaining and the rapid urease test (RUT), on gastric biopsy specimens obtained during gastrointestinal endoscopy were divided into 2 groups. Patients were allocated to one of the eradication regimens: triple therapy only or triple therapy combined with periodontal treatment. Each participant in both group received of a 10-day course of a proton pump inhibitor (Lansoprazole ) combined with amoxicillin (2 × 1 g daily) and clarithromycin (2 × 500 mg daily). Meanwhile, combined treatment group further received periodontal treatment consisted of scaling or combined with root planing and oral hygiene instructions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple therapy (Active Comparator): Conventional triple antibiotic treatment would be applied to all patients (consisted of a 10-day course of Lansoprazole (a proton pump inhibitor) combined with amoxicillin ( 2 × 1 g daily) and clarithromycin (2 × 500 mg daily).
  Interventions: Drug: Triple therapy
- Combined treatment (Experimental): Periodontal treatment would be administered in addition to triple therapy consisted of a 10-day course of a Lansoprazole (proton pump inhibitor )combined with amoxicillin (2 × 1 g daily) and clarithromycin (2 × 500 mg daily).
  Periodontal treatment consisted of supra and sub gingival scaling and root planing, oral hygiene instruction
  Interventions: Drug: Triple therapy; Procedure: professional periodontal treatment

INTERVENTIONS:
Drug: Triple therapy — triple therapy:a 10-day course of a Lansoprazole (proton pump inhibitor )combined with amoxicillin (2 × 1 g daily) and clarithromycin (2 × 500 mg daily).(trio)
  Other Names: Systemic eradication therapy
Procedure: professional periodontal treatment — periodontal treatment consisting of mechanical periodontal treatment (scaling and root planing) Oral hygiene insruction Periodontal treatment started concurrently with triple therapy
  Other Names: initial periodontal therapy
  Arms: Combined treatment

SUMMARY:
The efficacy of conventional systemic antibiotic therapy for eradication of gastric H. pylori has been seriously challenged by antibiotic resistance. Identification of alternative therapeutic strategies might help to overcome the limitation. The investigators' aim was to examine the effect of adjunct periodontal therapy, on gastric H. pylori eradication rate.

ELIGIBILITY:
Inclusion Criteria:

* tested positive for H. pylori both in gastric biopsy specimens and dental plaque samples

Exclusion Criteria:

The patients who had treatment with following medications within 6 months before the clinical protocol:

* had antibiotics
* had Proton pump inhibitor (PPI),
* had H2 blockers, and
* took bismuth derivatives
* had previous eradication therapy, or
* had previous periodontal therapy
* Edentulous patient
* Diabetic patients
* pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-04-21 (Actual); Primary Completion 2011-07-07 (Actual); Study Completion 2012-02-17 (Actual)

PRIMARY OUTCOMES:
eradication rate of gastric H. pylori infection | 3 months
  The follow-up was done by a 14C-urea breath test at least 12 weeks after completion of treatment . A 14C urea breath test analyzer (HUBT-20; Headway, Guangdong, China) was used to diagnose H. pylori infection

SECONDARY OUTCOMES:
oral H. pylori eradication | 3 months
  Oral H. pylori infection was tested by CLO test Plaque samples were collected from tooth surfaces with a sterile periodontal curette, then immediately inoculated onto CLO test gel.
periodontal parameters (Probing depth) | 3 months
  probing depth used as a surrogate marker to measure periodontal disease severity
Clinical Attachment level | 3 months
  used as a surrogate marker to measure severity of the periodontal disease
OHI (Oral Hygiene Index) | 3 months
  this index used to determine patient oral hygiene status (Greene and Vermillion, 1964)
Gingival Index | 3 months
  Löe-Silness gingival index
Plaque index | 3 months
  this index used to determine patient oral hygiene status (Silness-Löe)
Bleeding on Probing | 3 months
  an index give information on inflammation status of periodontal tissues

IPD SHARING:
Plan to Share IPD: Undecided